CLINICAL TRIAL: NCT02420353
Title: Evaluation of Recombinant Growth Hormone Therapy to Prevent Muscle Atrophy in Patients With Anterior Cruciate Ligament Tears
Brief Title: Evaluation of rGH Therapy to Prevent Muscle Atrophy in Patients With ACL Tears
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Christopher Mendias, PhD, ATC, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00087702; IND Exemption 123189 (Other: FDA)
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: muscle atrophy; growth hormone; ACL tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Muscular Atrophy | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Somatropin (Active Comparator): Somatropin of rDNA origin
  Interventions: Drug: Somatropin
- Placebo (Placebo Comparator): A placebo vehicle that contains somatropin diluent but no active hormone.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Somatropin — GH dose will be calculated by nomogram estimation of body surface area, and will be administered via subcutaneous injection in the abdominal area twice per day (BID) at a dose of 0.5mg GH per body surface area (BSA) in m2 (0.5mg/m2). Patients will begin GH treatment one week prior to surgery and will continue through 5 weeks after surgery. On the day of surgery, patients will not take GH, but otherwise patients will take GH every day over this 6 week period.
  Arms: Somatropin
Drug: Placebo — A placebo diluent that will be administered via subcutaneous injection in the abdominal area twice per day (BID) at a dose of the equivalent concentration of 0.5mg GH per body surface area (BSA) in m2 (0.5mg/m2). Patients will begin treatment one week prior to surgery and will continue through 5 weeks after surgery. On the day of surgery, patients will not take medication, but otherwise patients will take medication every day over this 6 week period.
  Arms: Placebo

SUMMARY:
Anterior cruciate ligament (ACL) tears are among the most frequent traumatic knee injuries that occur in physically active individuals. Despite advances in minimally invasive surgical reconstruction techniques and aggressive rehabilitation, this atrophy and loss of strength can persist even after patients return to full activity and can place them at considerable risk for re-injury and developing osteoarthritis (OA). The design of new therapeutic interventions to prevent muscle atrophy is needed to advance the care of patients who suffer from ACL injuries. The growth hormone (GH)/insulin-like growth factor-1 (IGF-1) axis plays an important role in promoting muscle growth and protecting muscle from atrophy. While GH therapy has shown promise in protecting immobilized muscle from various models of disuse atrophy, it remains unknown whether GH can help to restore strength and protect against the loss in strength that occurs after ACL tear. GH therapy may help to accelerate the safe return to play of patients that suffer ACL tears, and help to prevent the long-term OA and reduction in quality of life that occur after these traumatic knee injuries.

ELIGIBILITY:
Inclusion Criteria:

* Males between the ages of 18 and 35
* Have acute unilateral complete ACL tears with or without bucket handle medial meniscus tears that occurred within the past 6 months
* Consent to undergo an ACL reconstruction by an orthopaedic surgeon using a patellar tendon or hamstring autograft
* Will be performing supervised post-operative rehabilitation at UMHS MedSport at Dominos Farms

Exclusion Criteria:

* Patients who are undergoing a revision ACL reconstruction
* Had a previous injury to the involved knee
* Have an allergy to recombinant GH
* Have a BMI<20 or >35
* Have a growth disorder of bones or connective tissue, type 1 diabetes mellitus, type 2 diabetes mellitus, or who have a history of carpal tunnel syndrome, trigger finger, myopathy, cancer, endocrine disorder, hypertension or rheumatologic disorder.
* Systolic blood pressure >140mm Hg or diastolic blood pressure >90mm Hg, or with resting heart rate >110 BPM or <40 BPM at screening.
* Additionally, because GH is currently listed as a banned substance by the World Anti-Doping Agency (WADA), National Collegiate Athletics Association (NCAA) and most professional sports agencies, we will exclude patients who are current collegiate, professional or elite athletes.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Mendias, PhD, ATC, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Boesen AP, Dideriksen K, Couppe C, Magnusson SP, Schjerling P, Boesen M, Kjaer M, Langberg H. Tendon and skeletal muscle matrix gene expression and functional responses to immobilisation and rehabilitation in young males: effect of growth hormone administration. J Physiol. 2013 Dec 1;591(23):6039-52. doi: 10.1113/jphysiol.2013.261263. Epub 2013 Sep 30. PMID 24081158
- [Background] Surya S, Horowitz JF, Goldenberg N, Sakharova A, Harber M, Cornford AS, Symons K, Barkan AL. The pattern of growth hormone delivery to peripheral tissues determines insulin-like growth factor-1 and lipolytic responses in obese subjects. J Clin Endocrinol Metab. 2009 Aug;94(8):2828-34. doi: 10.1210/jc.2009-0638. Epub 2009 May 26. PMID 19470622
- [Background] Mendias CL, Lynch EB, Davis ME, Sibilsky Enselman ER, Harning JA, Dewolf PD, Makki TA, Bedi A. Changes in circulating biomarkers of muscle atrophy, inflammation, and cartilage turnover in patients undergoing anterior cruciate ligament reconstruction and rehabilitation. Am J Sports Med. 2013 Aug;41(8):1819-26. doi: 10.1177/0363546513490651. Epub 2013 Jun 5. PMID 23739685
- [Background] Gelato M, McNurlan M, Freedland E. Role of recombinant human growth hormone in HIV-associated wasting and cachexia: pathophysiology and rationale for treatment. Clin Ther. 2007 Nov;29(11):2269-88. doi: 10.1016/j.clinthera.2007.11.004. PMID 18158071
- [Derived] Mendias CL, Enselman ERS, Olszewski AM, Gumucio JP, Edon DL, Konnaris MA, Carpenter JE, Awan TM, Jacobson JA, Gagnier JJ, Barkan AL, Bedi A. The Use of Recombinant Human Growth Hormone to Protect Against Muscle Weakness in Patients Undergoing Anterior Cruciate Ligament Reconstruction: A Pilot, Randomized Placebo-Controlled Trial. Am J Sports Med. 2020 Jul;48(8):1916-1928. doi: 10.1177/0363546520920591. Epub 2020 May 26. PMID 32452208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment completed at the University of Michigan Sports Medicine Clinic
Period: Overall Study
Arm/Group | Somatropin | Placebo
Started | 10 | 10
Allocation to Intervention | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Of the 20 subjects who began the study, 19 were included in the baseline analysis. One subject who withdrew from the study was not included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Somatropin | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Isokinetic Knee Strength (Nm) [Mean (Standard Deviation); unit: Newton Meters]
  Absolute Isokinetic Flexion 60 dg/s Surgical | 74.7 (27.9) | 77.5 (11.4) | 76.0 (21.2)
  Absolute Isokinetic Extension 60 dg/s Surgical | 127.9 (46.7) | 124.7 (43.1) | 126.3 (43.8)

OUTCOME MEASURES:

1. Primary Outcome: Normative Isokinetic Knee Extension Strength, Measured in Newton Meters (Nm) at 26 Weeks Post-op
Description: Isokinetic knee flexion and extension strength measurements were obtained in a System 3 dynamometer (BioDex, Shirley, New York). Isokinetic measurements were performed at a speed of 60º/sec from a range of 0º to 90º of knee flexion. Normalized values were calculated by dividing the value from the injured limb by the value from the contralateral, uninjured leg prior to surgery. For each measurement, the highest force from a series of 5 repetitions was used.
Time Frame: at 26 wks post-op
Population: A total of 19 participants were analyzed for bilateral isokinetic knee strength using the BioDex system 3 results where recorded in newton meters (Nm).
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 0.881 [0.701 to 1.061] | 0.681 [0.532 to 0.83]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Mixed effect model; Test type: Other; p = 0.0498, Mixed Models Analysis

2. Secondary Outcome: Normative Isokinetic Extension (Nm) at Pre-op (Baseline)
Description: as for outcome 1
Time Frame: at pre-op (baseline)
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 0.746 [0.627 to 0.865] | 0.816 [0.651 to 0.981]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects model; p = 0.7024, Mixed Models Analysis

3. Secondary Outcome: Normative Isokinetic Flexion (Nm) at Pre-op (Baseline)
Description: as for outcome 1
Time Frame: at pre-op (baseline)
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 0.738 [0.643 to 0.833] | 0.92 [0.772 to 1.068]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects model; p = 0.135, Mixed Models Analysis

4. Secondary Outcome: Normative Isokinetic Flexion (Nm) at 26 Weeks Post-op
Description: as for outcome 1
Time Frame: at 26 weeks post-op
Population: A total of 19 participants were analyzed for bilateral isokinetic knee strength using the BioDex system 3 results where recorded in newton meters (Nm), results where then normalized to the participants nonsurgical limb.
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 1.068 [0.955 to 1.181] | 1.028 [0.841 to 1.215]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects model; p = 0.6836, Mixed Models Analysis

5. Secondary Outcome: Normative Isometric Extension (Nm) at Pre-op (Baseline)
Description: Isometric knee flexion and extension strength measurements were obtained in a System 3 dynamometer (BioDex, Shirley, New York). Isometric measurements were performed at 45º of knee flexion. Normalized values were calculated by dividing the value from the injured limb by the value from the contralateral, uninjured leg prior to surgery. For each measurement, the highest force from a series of 5 repetitions was used.
Time Frame: at pre-op (baseline)
Population: A total of 19 participants were analyzed for bilateral isometric knee strength using the BioDex system 3 results where recorded in newton meters (Nm).
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 0.761 [0.646 to 0.876] | 0.778 [0.676 to 0.88]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.9271, Mixed Models Analysis

6. Secondary Outcome: Normative Isometric Extension (Nm) at 26 Weeks Post-op
Description: as for outcome 5
Time Frame: at 26 weeks post-op
Population: as for outcome 4
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 0.718 [0.64 to 0.796] | 0.633 [0.513 to 0.753]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.1576, Mixed Models Analysis

7. Secondary Outcome: Normative Isometric Flexion (Nm) at Pre-op (Baseline)
Description: as for outcome 5
Time Frame: at pre-op (baseline)
Population: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 0.771 [0.641 to 0.901] | 0.867 [0.732 to 1.002]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.5586, Mixed Models Analysis

8. Secondary Outcome: Normative Isometric Flexion (Nm) at 26 Weeks Post-op
Description: as for outcome 5
Time Frame: at 26 weeks post-op
Population: as for outcome 4
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 1.017 [0.766 to 1.268] | 0.954 [0.847 to 1.061]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.45, Mixed Models Analysis

9. Secondary Outcome: Absolute Isokinetic Extension (Nm) at Pre-op (Baseline)
Description: Absolute Isokinetic knee flexion and extension strength measurements were obtained in a System 3 dynamometer (BioDex, Shirley, New York). Isokinetic measurements were performed at a speed of 60º/sec from a range of 0º to 90º of knee flexion. For each measurement, the highest force from a series of 5 repetitions was used.
Time Frame: at pre-op (baseline)
Population: A total of 19 participants were analyzed for bilateral isokinetic knee strength using the BioDex system 3 results where recorded in newton meters (Nm), results where then compared between study groups.
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 127.9 [100.8 to 155] | 124.7 [98 to 151.4]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.8573, Mixed Models Analysis

10. Secondary Outcome: Absolute Isokinetic Extension (Nm) at 26 wk Post-op
Description: Absolute Isokinetic knee flexion and extension strength measurements were obtained in a System 3 dynamometer (BioDex, Shirley, New York). Isokinetic measurements were performed at a speed of 60º/sec from a range of 0º to 90º of knee flexion. Strength values were calculated by comparing the affected limb of each subject across study group. For each measurement, the highest force from a series of 5 repetitions was used.
Time Frame: at 26 wk post-op
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 140.1 [111.7 to 168.5] | 105.6 [79.7 to 131.5]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.0564, Mixed Models Analysis

11. Secondary Outcome: Absolute Isokinetic Flexion (Nm) at Pre-op (Baseline)
Description: as for outcome 9
Time Frame: at pre-op (baseline)
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 74.7 [58.5 to 90.9] | 77.5 [70.4 to 84.6]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.7883, Mixed Models Analysis

12. Secondary Outcome: Absolute Isokinetic Flexion (Nm) at 26 Weeks Post-op
Description: as for outcome 10
Time Frame: at 26 weeks post-op
Population: A total of 19 participants were analyzed for bilateral isometric knee strength using the BioDex system 3 results where recorded in newton meters (Nm), results where then compared between study groups.
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 103.9 [85.3 to 122.5] | 86.2 [77.9 to 95.4]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.0901, Mixed Models Analysis

13. Secondary Outcome: Absolute Isometric Extension (Nm) at Pre-op (Baseline)
Description: Isometric knee flexion and extension strength measurements were obtained in a System 3 dynamometer (BioDex, Shirley, New York). Isometric measurements were performed at 45º of knee flexion. For each measurement, the highest force from a series of 5 repetitions was used.
Time Frame: at pre-op (baseline)
Population: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 183.1 [147.4 to 218.8] | 172.1 [139 to 205.2]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.6292, Mixed Models Analysis

14. Secondary Outcome: Absolute Isometric Extension (Nm) at 26 Weeks Post-op
Description: Absolute Isometric knee flexion and extension strength measurements were obtained in a System 3 dynamometer (BioDex, Shirley, New York). Isometric measurements were performed at 45º of knee flexion. Strength values were calculated by comparing the affected limb of each subject across study group. For each measurement, the highest force from a series of 5 repetitions was used.
Time Frame: at 26 weeks post-op
Population: as for outcome 12
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 172.4 [145.8 to 199] | 140.3 [107.4 to 173.2]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.161, Mixed Models Analysis

15. Secondary Outcome: Absolute Isometric Flexion (Nm) at Pre-op (Baseline)
Description: as for outcome 13
Time Frame: at pre-op (baseline)
Population: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 69.2 [55.7 to 82.7] | 77.2 [63.6 to 90.8]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.4437, Mixed Models Analysis

16. Secondary Outcome: Absolute Isometric Flexion (Nm) at 26 Weeks Post-op
Description: as for outcome 14
Time Frame: at 26 weeks post-op
Population: as for outcome 12
Measure: Mean (90% Confidence Interval); unit: Nm
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Nm | 84.6 [74 to 95.2] | 88.1 [72.4 to 103.8]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.7325, Mixed Models Analysis

17. Secondary Outcome: VR12 Health Survey: Physical Health Summary Measure Score at Pre-op (Baseline)
Description: The VR-12 includes 12 questions that do not give an overall score but yield a physical and mental component score. PCS and MCS summary scores are standardized using a t-score transformation and normalized to the U.S. population of a score of 50 and a standard deviation of 10. Higher PCS and MCS scores indicate better health. Medical Expenditure Panel Survey (MEPS) collected between 2000 and 2002 standard norms range as followed PCS maximum: 72.11; minimum: 0.59.
Time Frame: at pre-op (baseline)
Population: A total of 19 participants were administered the VR12 survey, this 12 part questionnaire is then score in two parts based on the answers selected by the subjects.
Measure: Mean (90% Confidence Interval); unit: T-score
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
T-score | 46.5 [40.9 to 52.1] | 45.1 [40.6 to 49.6]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects analysis; p = 0.6291, Mixed Models Analysis

18. Secondary Outcome: VR12 Health Survey: Physical Health Summary Measure Score at 26 Weeks Post-op
Description: as for outcome 17
Time Frame: at 26 weeks post-op
Population: as for outcome 17
Measure: Mean (90% Confidence Interval); unit: T-score
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
T-score | 52.9 [51.2 to 54.6] | 50.2 [47.6 to 52.8]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed-effects model; p = 0.3332, Mixed Models Analysis

19. Secondary Outcome: VR12 Health Survey: Mental Health Summary Measure Score at Pre-op (Baseline)
Description: The VR-12 includes 12 questions that do not give an overall score but yield a physical and mental component score. PCS and MCS summary scores are standardized using a t-score transformation and normalized to the U.S. population of a score of 50 and a standard deviation of 10. Higher PCS and MCS scores indicate better health. Medical Expenditure Panel Survey (MEPS) collected between 2000 and 2002 standard norms range as followed MCS Maximum: 76.09; Minimum: -2.47.
Time Frame: at pre-op (baseline)
Population: as for outcome 17
Measure: Mean (90% Confidence Interval); unit: T-score
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
T-score | 54.6 [48.8 to 60.4] | 55.6 [51.7 to 59.5]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects analysis; p = 0.79, Mixed Models Analysis

20. Secondary Outcome: VR12 Health Survey: Mental Health Summary Measure Score at 26 Weeks Post-op
Description: as for outcome 19
Time Frame: at 26 weeks post-op
Population: as for outcome 17
Measure: Mean (90% Confidence Interval); unit: T-score
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
T-score | 56.7 [52.9 to 60.5] | 59.3 [56.3 to 62.3]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects analysis; p = 0.4965, Mixed Models Analysis

21. Secondary Outcome: International Knee Document Committee (IKDC) at Pre-op (Baseline)
Description: The IKDC percentage score is a subjective patients reported outcome measure (PROM) that scores a participants over all score. The PROM looks at 3 categories: symptoms, sports activity, and knee function. Scores range from 0 to 100, the final score given is interpreted as a measure of function with higher scores representing higher levels of function.
Time Frame: at pre-op (baseline)
Population: A total of 19 participants complete the IKDC outcome measure, the form was administer by hand at the time of the study visits for each study timepoint.
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 54.6 [48.8 to 60.4] | 55.6 [51.7 to 59.5]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects analysis; p = 0.1331, Mixed Models Analysis

22. Secondary Outcome: International Knee Documentation Committee (IKDC) up to 26 wk Post-op
Description: as for outcome 21
Time Frame: up to 26 wk post-op
Population: as for outcome 21
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale | 65 [60.6 to 69.4] | 67 [58.7 to 75.3]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed-model analysis; p = 0.5251, Mixed Models Analysis

23. Secondary Outcome: The Knee Injury and Osteoarthritis Outcome Score (KOOS): Patient Reported Outcome Measure: ADL at 26 Weeks Post-op
Description: KOOS Function in daily living (ADL) (17 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. An aggregate total score is not calculated since it is regarded desirable to analyze and interpret the five dimensions separately.
  Maximum score 100% / Minimum score 0%. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures
Time Frame: at 26 weeks post-op
Population: A total of 19 participants were administered the KOOS survey, this 42 part questionnaire is then score in five parts based on the answers selected by the subjects.
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 98 [96 to 100] | 98.0 [95.6 to 100.4]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects analysis; p = 0.1064, Mixed Models Analysis

24. Secondary Outcome: KOOS Patient Reported Outcome Measure: ADL at Pre-op (Baseline)
Description: as for outcome 23
Time Frame: at pre-op (baseline)
Population: as for outcome 23
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 88 [82.8 to 93.2] | 91 [84.1 to 97.9]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects analysis; p = 0.4852, Mixed Models Analysis

25. Secondary Outcome: KOOS Patient Reported Outcome Measure: Pain at 26 Weeks Post-op
Description: KOOS Pain (9 items) A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. An aggregate total score is not calculated since it is regarded desirable to analyze and interpret the five dimensions separately.
  Maximum score 100% / Minimum score 0%. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures
Time Frame: at 26 weeks post-op
Population: as for outcome 23
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 91 [88.1 to 93.9] | 92 [87.2 to 96.8]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other; p = 0.7943, Mixed Models Analysis

26. Secondary Outcome: KOOS Patient Reported Outcome Measure: Pain at Pre-op (Baseline)
Description: as for outcome 25
Time Frame: at pre-op (baseline)
Population: as for outcome 23
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 74 [69.2 to 78.8] | 83 [75 to 91]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other; p = 0.0894, Mixed Models Analysis

27. Secondary Outcome: KOOS Patient Reported Outcome Measure: Quality of Life at 26 Weeks Post-op
Description: KOOS Quality of Life (QoL) (4 items) A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. An aggregate total score is not calculated since it is regarded desirable to analyze and interpret the five dimensions separately.
  Maximum score 100% / Minimum score 0%. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures
Time Frame: at 26 weeks post-op
Population: as for outcome 23
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 53 [42.8 to 63.2] | 63 [53.1 to 72.9]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects analysis; p = 0.0673, Mixed Models Analysis

28. Secondary Outcome: KOOS Patient Reported Outcome Measure: Quality of Life at Pre-op (Baseline)
Description: as for outcome 27
Time Frame: at pre-op (baseline)
Population: as for outcome 23
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 33 [23.1 to 42.9] | 47 [31.1 to 62.9]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects analysis; p = 0.0185, Mixed Models Analysis

29. Secondary Outcome: KOOS Patient Reported Outcome Measure: Sport and Recreation at 26 Weeks Post-op
Description: KOOS Sport and Recreation (Sport/Rec) (5 items) A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. An aggregate total score is not calculated since it is regarded desirable to analyze and interpret the five dimensions separately.
  Maximum score 100% / Minimum score 0%. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures.
Time Frame: at 26 weeks post-op
Population: as for outcome 23
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 67.5 [57.3 to 77.7] | 72.2 [56.2 to 88.2]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects analysis; p = 0.6094, Mixed Models Analysis

30. Secondary Outcome: KOOS Patient Reported Outcome Measure: Sports and Recreation at Pre-op (Baseline)
Description: as for outcome 29
Time Frame: at pre-op (baseline)
Population: as for outcome 23
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 46.5 [30.7 to 62.3] | 55.6 [41.1 to 70.1]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects analysis; p = 0.3279, Mixed Models Analysis

31. Secondary Outcome: KOOS Patient Reported Outcome Measure: Symptoms at 26 Weeks Post-op
Description: KOOS Symptoms (7 items) A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. An aggregate total score is not calculated since it is regarded desirable to analyze and interpret the five dimensions separately.
  Maximum score 100% / Minimum score 0%. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures
Time Frame: at 26 weeks post-op
Population: as for outcome 23
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 60 [52.9 to 67.1] | 68 [62.8 to 73.2]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects analysis; p = 0.2802, Mixed Models Analysis

32. Secondary Outcome: KOOS Patient Reported Outcome Measure: Symptoms at Pre-op (Baseline)
Description: as for outcome 31
Time Frame: at pre-op (baseline)
Population: as for outcome 23
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | 53 [45.7 to 60.3] | 64 [59.9 to 68.1]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other; p = 0.1064, Mixed Models Analysis

33. Secondary Outcome: Absolute Quadriceps Volume (L) at Pre-op (Baseline)
Description: Bilateral MRI scans were obtained at specific time points to assess the muscle volume of the quadriceps and hamstring muscle groups will be calculated using GE ImagePACS software (FDA cleared software which is the standard software used to read and analyze imaging studies in the UMHS).
Time Frame: at pre-op (baseline)
Population: Scans were performed on a total of 19 participant at three time points throughout the study.
Measure: Mean (90% Confidence Interval); unit: Liters
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Liters | 2.48 [2.16 to 2.8] | 2.12 [1.97 to 2.27]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.0509, Mixed Models Analysis

34. Secondary Outcome: Absolute Quadricep Volume (L) at 26 Week Post-op
Description: as for outcome 33
Time Frame: at 26 week post-op
Population: Scans were performed on a total of 19 participant at three time points throughout the study.
Measure: Mean (90% Confidence Interval); unit: Liters
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Liters | 2.27 [2.02 to 2.52] | 2.12 [1.88 to 2.36]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects analysis; p = 0.1605, Mixed Models Analysis

35. Secondary Outcome: Absolute Hamstring Volume (L) at Pre-op (Baseline)
Description: as for outcome 33
Time Frame: at pre-op (baseline)
Population: Scans were performed on a total of 19 participant at three time points throughout the study.
Measure: Mean (90% Confidence Interval); unit: Liters
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Liters | 1 [0.93 to 1.07] | 0.88 [0.85 to 0.91]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.0357, Mixed Models Analysis

36. Secondary Outcome: Absolute Hamstring Volume (L) at 26 Weeks Post-op
Description: as for outcome 33
Time Frame: at 26 weeks post-op
Population: Scans were performed on a total of 19 participant at three time points throughout the study.
Measure: Mean (90% Confidence Interval); unit: Liters
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Liters | 0.98 [0.89 to 1.07] | 0.88 [0.84 to 0.92]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.0122, Mixed Models Analysis

37. Secondary Outcome: Normalized Quadriceps Volume (L) at Pre-op (Baseline)
Description: Normalized volume relative to the pre-op measurements of the uninjured limb, used to assess the muscle volume of the quadriceps and hamstring muscle groups will be calculated using GE ImagePACS software (FDA cleared software which is the standard software used to read and analyze imaging studies in the UMHS).
Time Frame: at pre-op (baseline)
Population: Scans were performed on a total of 19 participant at three time points throughout the study.
Measure: Mean (90% Confidence Interval); unit: Liters
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Liters | 1 [0.87 to 1.13] | 0.85 [0.79 to 0.91]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.5853, Mixed Models Analysis

38. Secondary Outcome: Normalized Quadriceps Volume (L) at 26 Weeks Post-op
Description: as for outcome 37
Time Frame: at 26 weeks post-op
Population: Scans were performed on a total of 19 participant at three time points throughout the study.
Measure: Mean (90% Confidence Interval); unit: Liters
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Liters | 0.91 [0.81 to 1.01] | 0.85 [0.75 to 0.95]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.6288, Mixed Models Analysis

39. Secondary Outcome: Normalized Hamstring Volume (L) at Pre-op (Baseline)
Description: as for outcome 37
Time Frame: at pre-op (baseline)
Population: Scans were performed on a total of 19 participant at three time points throughout the study.
Measure: Mean (90% Confidence Interval); unit: Liters
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Liters | 1.06 [0.99 to 1.13] | 0.93 [0.89 to 0.97]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.5022, Mixed Models Analysis

40. Secondary Outcome: Normalized Hamstring Volume (L) at 26 Weeks Post-op
Description: as for outcome 37
Time Frame: at 26 weeks post-op
Population: Scans were performed on a total of 19 participant at three time points throughout the study.
Measure: Mean (90% Confidence Interval); unit: Liters
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
Liters | 1.03 [0.94 to 1.12] | 0.93 [0.88 to 0.98]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.7507, Mixed Models Analysis

41. Secondary Outcome: Insulin Like Growth Factor (IGF1) at -1 and 5 Weeks Post-op
Description: IGF1 was measured from serum using an IMMULITE 2000 system (Siemens).
Time Frame: Area under the curve between -1 and 5 weeks post-op
Population: Blood was drawn from the antecubital vein from each patient at specific time points, plasma and serum were prepared from whole blood and stored at -80ºC.
Measure: Mean (90% Confidence Interval); unit: ng*days/mL
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
ng*days/mL | 22478 [19505 to 25451] | 10626 [8749 to 12503]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p < .0001, Mixed Models Analysis

42. Secondary Outcome: Myostatin at -1 and 5 Weeks Post-op
Description: Myostatin was measured from plasma using ELISAs (R&D Systems, Minneapolis, MN) following manufacturer recommendations.
Time Frame: Area under the curve between -1 and 5 weeks post-op
Population: as for outcome 41
Measure: Mean (90% Confidence Interval); unit: ng*days/mL
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
ng*days/mL | 190.7 [170.3 to 211.1] | 193.6 [175.3 to 211.9]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.8581, Mixed Models Analysis

43. Secondary Outcome: MMP3 at -1 and 5 Weeks Post-op
Description: Matrix metalloproteinase-3 (MMP3) was measured from serum using ELISAs (R&D Systems, Minneapolis, MN) following manufacturer recommendations.
Time Frame: Area under the curve between -1 and 5 weeks post-op
Population: as for outcome 41
Measure: Mean (90% Confidence Interval); unit: ng*days/mL
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
ng*days/mL | 1188 [924 to 1452] | 766 [631 to 901]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — mixed effects model; p = 0.0208, Mixed Models Analysis

44. Secondary Outcome: Hyaluronic Acid at -1 and 5 Weeks Post-op
Description: Hyaluronic acid was measured from plasma using ELISAs (R&D Systems, Minneapolis, MN) following manufacturer recommendations.
Time Frame: Area under the curve between -1 and 5 weeks post-op
Population: as for outcome 41
Measure: Mean (90% Confidence Interval); unit: ng*days/mL
Arm/Group | Somatropin | Placebo
Number analyzed (Participants) | 10 | 9
ng*days/mL | 190.7 [170.3 to 211.1] | 193.6 [175.3 to 211.9]
Statistical Analysis 1: Comparison: Somatropin vs Placebo; Test type: Other — Mixed effects model; p = 0.8581, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1-3 weeks pre-op to 25 weeks post-op
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Somatropin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 5/10 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatropin (N=10) | Placebo (N=9)
Back pain (General disorders) | 5 (5) | 5 (5)
Fatigue (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Joint pain (other than surgical knee) (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Headache (General disorders) | 3 (3) | 3 (3)
Increased sweating (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Tingling sensation/numbness (General disorders) | 2 (2) | 1 (1)
Elevated alanine aminotransferase (General disorders) | 2 (2) | 3 (3)
Elevated aspirate aminotransferase (General disorders) | 2 (2) | 3 (3)
Temperature sensation fluctuations (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Reduced appetite (General disorders) | 1 (1) | 0 (0)
Elevated blood glucose (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Muscle spasms/cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Please consult the full manuscript or contact the study PI for any questions about study results. Additional clinical trials must be conducted before definitive conclusions can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT02420353/Prot_SAP_000.pdf